CLINICAL TRIAL: NCT02820064
Title: Effects of Hypoxia and Inflammation on Citrulline Synthesis by Ornithine Transcarbamylase in Human Enterocytes
Acronym: HYPOCITRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC15.303
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Hypoxia; Inflammation; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Hypoxia; Inflammation; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- only one arm (Other): Patients for who and esophagogastroduodenoscopy in order to diagnose is performed. 8 duodenal biopsy specimens will be removed.
  Interventions: Procedure: duodenal biopsy during gastroduodenal endoscopy

INTERVENTIONS:
Procedure: duodenal biopsy during gastroduodenal endoscopy — Patients for who and esophagogastroduodenoscopy in order to diagnose is performed. 8 duodenal biopsy specimens will be removed.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by chronic systemic hypoxia and low-grade inflammation as well as by an alteration of arginine (ARG) metabolism. As ARG is synthetized from circulating citrulline (CIT), an alteration of CIT homeostasis, particularly its production by ornithine transcarbamylase (OCT) in small intestine could be involved. We hypothesized that hypoxia +/- inflammation, classically associated to COPD, has effects on OCT regulation in enterocytes.

This study aims at exploring the effects of hypoxia and inflammation on the production of citrulline by ornithine transcarbamylase (OTC) activity in enterocytes from explant cultures of duodenal tissue.

DETAILED DESCRIPTION:
Citrulline is an amino-acid almost exclusively released by the small intestine after its synthesis from glutamine by the OTC in enterocytes. Citrulline from the small intestine is released into the portal vena and, because it does not enter hepatocytes, it reaches the systemic circulation to be metabolized in arginine by kidneys. By this way, is an important source of endogenous ARG. Moreover, evidence suggests that circulating citrulline could have a direct action on the regulation of muscle protein synthesis. Therefore, the administration of citrulline might be an interesting nutritional strategy to preserve or restore muscle mass and function. Muscle mass is a determinant of respiratory function and muscle weakness explains for a large part morbidity and mortality in patients suffering from Chronic Obstructive Pulmonary Disease (COPD).

Evidence suggests that citrulline plasmatic levels would be lower in several states involving systemic inflammation and hypoxia. Indeed, it has been observed in rats that hypoxia leads to a sharp decline in plasma CIT concentration and also in human (hypocitrullinemia has been observed in Intensive Care Unit patients and in subjects suffering from sepsis and trauma) but the cause of relationship is not yet established. Therefore, it may be supposed that a decreased plasma CIT level could be responsible for a decrease in de novo ARG synthesis leading to an impairment of NO production (endothelial dysfunction) in these pathological situations.

Because chronic hypoxia and systemic inflammation are both systemic traits of patients suffering from COPD, the fact that hypoxia and/or systemic inflammation might directly affect OCT, decreasing intestinal citrulline production which, in turn, could contribute to endothelial dysfunction and muscle weakness is considered.

In order to explore this hypothesis, the potential consequences of hypoxia and inflammation (alone or in association) on citrulline synthesis by the OCT in human enterocytes will be determined, thanks to an "explant" culture model of duodenal tissue. Duodenal biopsies will be removed during oesophago-gastro-duodenoscopies performed in the Hepato-gastro-enterology unit of Grenoble University Hospital, among patients expected to undergo a gastroscopy for any diagnostic purpose. 30 patients will be selected during a period of 6 months. After complete information and written agreement, 8 biopsy specimens will be removed from the duodenum of each patient and processed for organ culture.

Then, duodenal biopsies will be incubated in the presence or not of cytokines and exposed or not to hypoxia. Indeed, 4 groups will be constituted: a control group (no stimulus), a group exposed to hypoxic conditions, a group exposed to inflammatory conditions (cytokines) and a group exposed to both hypoxic an inflammatory conditions.

As primary endpoint, for each group, the OTC activity and the citrulline production in the culture medium will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Digestive disease known or suspected which justify an oeso-gastro-endoscopy with digestive biopsies, excepted a disease with duodenal localization known or strongly suspected.
* Gastroscopy performed under general anaesthesia
* Patient's written agreement obtained

Non inclusion-criteria:

* Age < 18
* Therapeutical endoscopy (that is to say when a therapeutical act will be performed as balloon dilation, digestive or biliary prosthesis, drainage, diverticulotomy, polypectomy, variceal ligation...) either expected or
* Duodenal pathology (known or strongly suspected with the clinical and biological elements)
* Duodenal biopsies are not allowed to be performed: vascular lesions, digestive haemorrhage, clotting disorder.
* Antiplatelet drug and anticoagulant drug
* Lack of written agreement
* Subjects hospitalized in an emergency state or without agreement
* Subjects who cannot be contacted in emergency.

Exclusion criteria:

subjects will be excluded from the study:

* if an unexpected therapeutic act has to be performed during the endoscopy
* if duodenal duodenal atrophy or lesions are discovered during the endoscopy
* if duodenal lesions are discoverd at the histological examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
OCT activity in biopsy specimens | OCT activity in biopsies after incubation
  OCT activity in duodenal biopsy specimens will be measured at the end of the incubation period and compared between the 4 different groups (standard/inflammatory/hypoxic:inflammatory+hypoxic conditions)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Fontaine, Professor, Principal Investigator — Division of clinical Nutrition-Grenoble University Hospital
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moinard C, Cynober L. Citrulline: a new player in the control of nitrogen homeostasis. J Nutr. 2007 Jun;137(6 Suppl 2):1621S-1625S. doi: 10.1093/jn/137.6.1621S. PMID 17513438
- [Background] Windmueller HG, Spaeth AE. Source and fate of circulating citrulline. Am J Physiol. 1981 Dec;241(6):E473-80. doi: 10.1152/ajpendo.1981.241.6.E473. PMID 7325229
- [Background] Breuillard C, Cynober L, Moinard C. Citrulline and nitrogen homeostasis: an overview. Amino Acids. 2015 Apr;47(4):685-91. doi: 10.1007/s00726-015-1932-2. Epub 2015 Feb 13. PMID 25676932
- [Background] Osowska S, Moinard C, Neveux N, Loi C, Cynober L. Citrulline increases arginine pools and restores nitrogen balance after massive intestinal resection. Gut. 2004 Dec;53(12):1781-6. doi: 10.1136/gut.2004.042317. PMID 15542514
- [Background] Osowska S, Duchemann T, Walrand S, Paillard A, Boirie Y, Cynober L, Moinard C. Citrulline modulates muscle protein metabolism in old malnourished rats. Am J Physiol Endocrinol Metab. 2006 Sep;291(3):E582-6. doi: 10.1152/ajpendo.00398.2005. Epub 2006 Apr 11. PMID 16608884
- [Background] Faure C, Raynaud-Simon A, Ferry A, Dauge V, Cynober L, Aussel C, Moinard C. Leucine and citrulline modulate muscle function in malnourished aged rats. Amino Acids. 2012 Apr;42(4):1425-33. doi: 10.1007/s00726-011-0841-2. Epub 2011 Feb 23. PMID 21344178
- [Background] Faure C, Morio B, Chafey P, Le Plenier S, Noirez P, Randrianarison-Huetz V, Cynober L, Aussel C, Moinard C. Citrulline enhances myofibrillar constituents expression of skeletal muscle and induces a switch in muscle energy metabolism in malnourished aged rats. Proteomics. 2013 Jul;13(14):2191-201. doi: 10.1002/pmic.201200262. Epub 2013 Jun 10. PMID 23592530
- [Background] Ventura G, Noirez P, Breuille D, Godin JP, Pinaud S, Cleroux M, Choisy C, Le Plenier S, Bastic V, Neveux N, Cynober L, Moinard C. Effect of citrulline on muscle functions during moderate dietary restriction in healthy adult rats. Amino Acids. 2013 Nov;45(5):1123-31. doi: 10.1007/s00726-013-1564-3. Epub 2013 Aug 3. PMID 23913268
- [Background] The economic burden of lung disease. European white lung book 2013:16-27.
- [Background] Antonione R. Nutrition in cardiac and pulmonary disease. In Basic in clinical nutrition. Sobotka L. ed. Galen, 4th ed. 485-493.
- [Background] Jonker R. and al. Whole body de novo ARG production and NO synthesis are reduced in COPD patients. Clin.Nutr. 2013;32(S1):S5-S6.
- [Background] Coeffier M, Miralles-Barrachina O, Le Pessot F, Lalaude O, Daveau M, Lavoinne A, Lerebours E, Dechelotte P. Influence of glutamine on cytokine production by human gut in vitro. Cytokine. 2001 Feb 7;13(3):148-54. doi: 10.1006/cyto.2000.0813. PMID 11161457
- [Background] Lecleire S, Coeffier M, Leblond J, Hubert A, Lemoulan S, Petit A, Ducrotte P, Dechelotte P, Marion R. Modulation of nitric oxide and cytokines production by L-arginine in human gut mucosa. Clin Nutr. 2005 Jun;24(3):353-9. doi: 10.1016/j.clnu.2004.11.011. PMID 15896421
- [Background] Hubert-Buron A, Leblond J, Jacquot A, Ducrotte P, Dechelotte P, Coeffier M. Glutamine pretreatment reduces IL-8 production in human intestinal epithelial cells by limiting IkappaBalpha ubiquitination. J Nutr. 2006 Jun;136(6):1461-5. doi: 10.1093/jn/136.6.1461. PMID 16702304
- [Background] Reimund JM, Wittersheim C, Dumont S, Muller CD, Kenney JS, Baumann R, Poindron P, Duclos B. Increased production of tumour necrosis factor-alpha interleukin-1 beta, and interleukin-6 by morphologically normal intestinal biopsies from patients with Crohn's disease. Gut. 1996 Nov;39(5):684-9. doi: 10.1136/gut.39.5.684. PMID 9026483
- [Background] Chan MF. Complications of upper gastrointestinal endoscopy. Gastrointest Endosc Clin N Am. 1996 Apr;6(2):287-303. PMID 8673329
- [Background] Christensen M, Achiam M, Trap R, Stockel M, Rosenberg J, Schulze S. Transnasal gastroscopy. Dan Med Bull. 2000 Jun;47(3):218-20. PMID 10913986
- [Background] Zubarik R, Eisen G, Mastropietro C, Lopez J, Carroll J, Benjamin S, Fleischer DE. Prospective analysis of complications 30 days after outpatient upper endoscopy. Am J Gastroenterol. 1999 Jun;94(6):1539-45. doi: 10.1111/j.1572-0241.1999.01141.x. PMID 10364022
- [Background] Dumortier J, Ponchon T, Scoazec JY, Moulinier B, Zarka F, Paliard P, Lambert R. Prospective evaluation of transnasal esophagogastroduodenoscopy: feasibility and study on performance and tolerance. Gastrointest Endosc. 1999 Mar;49(3 Pt 1):285-91. doi: 10.1016/s0016-5107(99)70002-7. PMID 10049409
- [Background] Lacy PD, Lee JM, O'Morain CA. Temporomandibular joint dislocation: an unusual complication of upper gastrointestinal endoscopy. Am J Gastroenterol. 2000 Dec;95(12):3653-4. doi: 10.1111/j.1572-0241.2000.03396.x. No abstract available. PMID 11151916
- [Background] Kise Y, Suzuki R, Shimada H, Tanaka H, Oshiba G, Chino O, Makuuchi H. Idiopathic submucosal hematoma of esophagus complicated by dissecting aneurysm, followed-up endoscopically during conservative treatment. Endoscopy. 2001 Apr;33(4):374-8. doi: 10.1055/s-2001-13684. PMID 11315902
- [Background] Vu CK, Korman MG, Bejer I, Davis S. Gastrointestinal bleeding after cold biopsy. Am J Gastroenterol. 1998 Jul;93(7):1141-3. doi: 10.1111/j.1572-0241.1998.346_e.x. PMID 9672346
- [Background] Giudicelli R. [Esophageal perforations. Results of a national survey]. Ann Chir. 1992;46(2):183-7. No abstract available. French. PMID 1605545
- [Background] Giangreco E, D'agate C, Barbera C, Puzzo L, Aprile G, Naso P, Bonanno G, Russo FP, Nicoletti A, Incarbone S, Trama G, Russo A. Prevalence of celiac disease in adult patients with refractory functional dyspepsia: value of routine duodenal biopsy. World J Gastroenterol. 2008 Dec 7;14(45):6948-53. doi: 10.3748/wjg.14.6948. PMID 19058330
- [Background] Heresbach D, Napoléon B. Delchier J.C. and al. Consensus en endoscopie digestive. Acta endo (2009) 39 :206-2011.
- [Background] Prat F. Recommandations de la SFED 2005 : De la pratique des biopsies oeso-gastro-duodénales.
- [Background] Boustière C. Endoscopie digestive, antigoagulants, antiagrégants : faut-il encore modifier nos pratiques en 2013 ? Acta endo (2013) 43 :260-265.
- [Background] Boustiere C, Veitch A, Vanbiervliet G, Bulois P, Deprez P, Laquiere A, Laugier R, Lesur G, Mosler P, Nalet B, Napoleon B, Rembacken B, Ajzenberg N, Collet JP, Baron T, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Endoscopy and antiplatelet agents. European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2011 May;43(5):445-61. doi: 10.1055/s-0030-1256317. Epub 2011 May 4. PMID 21547880
- [Background] Recommandations de bonnes pratiques sur les antiagrégants plaquettaires: prise en compte des risques thrombotique et hémorragique en cas de geste endoscopique HAS-SFED, oct 2012.
- [Background] Napoleon B, Boneu B, Maillard L, Samama CM, Schved JF, Gay G, Ponchon T, Sautereau D, Canard JM; Board of the French Society for Digestive Endoscopy (SFED). Guidelines of the French Society for Digestive Endoscopy (SFED). Endoscopy. 2006 Jun;38(6):632-8. doi: 10.1055/s-2006-925086. Epub 2006 Mar 14. No abstract available. PMID 16586249
- [Background] Ventura G, Moinard C, Sinico F, Carriere V, Lasserre V, Cynober L, De Bandt JP. Evidence for a role of the ileum in the control of nitrogen homeostasis via the regulation of arginine metabolism. Br J Nutr. 2011 Jul;106(2):227-36. doi: 10.1017/S0007114511000079. PMID 22568979